CLINICAL TRIAL: NCT04103385
Title: Reconnecting: Improving Interoception to Reduce Suicidal Ideation in the Military
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miami University (Other)
Collaborators: Auburn University (Other)
Responsible Party: Principal Investigator, April Smith, Assistant Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G03177
Record Dates: First submitted 2019-09-19; First posted 2019-09-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Suicidal Ideation; Interoception
Keywords: interoception; suicidal ideation; suicide; military; intervention; clinical trial
MeSH Terms: conditions — Suicidal Ideation; Suicide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: We will attempt to mask care provider. The Investigators will be completely blind to condition assignment. Outcomes will be assessed via computer and thus will also be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reconnecting to Internal Sensations and Experiences (Experimental): Aims to improve "interoception" or connection to the body's emotions & internal sensation and reduce suicidal ideation.
  Interventions: Behavioral: RISE (Reconnecting to Internal Sensations and Experiences)
- Restoring Individual Strength and Energy (Active Comparator): Aims to reduce life stressors and improve physical health
  Interventions: Behavioral: RISE (Reconnecting to Individual Strength and Energy)

INTERVENTIONS:
Behavioral: RISE (Reconnecting to Internal Sensations and Experiences) — The overarching goal of RISE is to increase interoception by reconnecting people with their internal sensations
  Arms: Reconnecting to Internal Sensations and Experiences
Behavioral: RISE (Reconnecting to Individual Strength and Energy) — Aims to reduce life stressors and improve physical health
  Arms: Restoring Individual Strength and Energy

SUMMARY:
Background: Interoception is defined as the "sense of the physiological condition of the entire body" and is crucial for recognizing emotions and sensations (e.g., hunger, temperature, pain) and responding accordingly. The investigator's lab has conducted several independent studies and two pilot studies that support the hypothesis that disrupted interoception leads one to be disconnected from the body, and thus more able to harm the body should one desire to do so. Research suggests that interoceptive deficits may not only differentiate those who are thinking about suicide from those who engage in suicidal behavior, but it may also provide information about who is at imminent risk for suicidal behavior. The identification of novel, short-term risk factors, like interoceptive deficits, allows for the development of new treatment applications for suicide, which is important for several reasons: 1) suicide rates have increased in recent years, especially among military populations, and 2) existing treatment approaches are often ineffective, lengthy, expensive, or impractical for large-scale dissemination. This project evaluates a novel, brief intervention for interoceptive deficits and suicidal behavior with the potential to be acceptable and feasible for a military population.

DETAILED DESCRIPTION:
Background: Interoception is defined as the "sense of the physiological condition of the entire body" and is crucial for recognizing emotions and sensations (e.g., hunger, temperature, pain) and responding accordingly. The investigator's lab has conducted several independent studies and two pilot studies that support the hypothesis that disrupted interoception leads one to be disconnected from the body, and thus more able to harm the body should one desire to do so. Research suggests that interoceptive deficits may not only differentiate those who are thinking about suicide from those who engage in suicidal behavior, but it may also provide information about who is at imminent risk for suicidal behavior. The identification of novel, short-term risk factors, like interoceptive deficits, allows for the development of new treatment applications for suicide, which is important for several reasons: 1) suicide rates have increased in recent years, especially among military populations, and 2) existing treatment approaches are often ineffective, lengthy, expensive, or impractical for large-scale dissemination. This project evaluates a novel, brief intervention for interoceptive deficits and suicidal behavior with the potential to be acceptable and feasible for a military population.

Specific Aims and Hypotheses:

Aim 1: Determine whether the interoception training procedure (Reconnecting to Internal Sensations and Experiences [RISE]) decreases interoceptive deficits, suicidal ideation compared to a control condition. H1: Participants receiving the interoceptive training will demonstrate decreased interoceptive deficits relative to controls and relative to their pre-training levels.

H2: Participants receiving the interoceptive training will demonstrate decreased suicidal ideation relative to controls and relative to their pre-training levels.

H3: Group differences between the interoceptive training and control conditions will be maintained at one- and three-month follow-ups.

Aim 2: Establish the feasibility and acceptability of the RISE intervention in a military sample.

H4: Participants and clinic personnel will find the intervention to be feasible and acceptable.

Study Design: Potential participants will be recruited from military bases' IOPs. Eligible participants will be invited to complete the baseline assessment and will be assigned to one of two conditions: 1) RISE, or 2) control (reading health related material). Participants in the RISE condition will complete four 45-minute online sessions of training that focus on multiple aspects of interoception including: body awareness, body sensations and movement, eating, health and self-care, emotional awareness, and understanding the self in relation to others. Outcome assessments will be administered at post-treatment and at one- and three-month-follow-ups.

Due to the COVID-19 pandemic, which temporarily paused data collection at two of the study sites (Wright Patterson Medical Center & Madigan Army Medical Center), a fully online arm of the study was added in June 2020. Data collection was later able to be resumed at all study sites. When we added this fully arm, we increased our planned recruitment goal from 132 to 200. Data collection was ultimately concluded with an enrolled N of 195.

Military Benefit: Interoceptive deficits are an important treatment target for military personnel for several reasons. First, experiences particular to military populations (e.g., stress, trauma) are believed to lead to interoceptive deficits. Second, the broad construct of interoceptive deficits and the individual components of interoceptive deficits are related to suicidal ideation and behavior among Service members. Third, our research finds that interoceptive deficits are easily modifiable, and that increasing interoception reduces risk factors for suicide. Fourth, the entire intervention can be delivered electronically and is brief, which allows it to circumvent barriers to treatment associated with traditional face-to-face therapy. Fifth, because of its portability, the intervention can be provided to deployed Service members and it can be delivered as a standalone intervention or as an add-on to existing treatments. In sum, our proposed intervention has implications not only for the reduction of suicidal behavior, but also for improvements in military performance and future functioning.

ELIGIBILITY:
Inclusion Criteria:

* Being seen for behavioral health services at Wright-Patterson Medical Center (WPMC) or Madigan Army Medical Center (MAMC) for participants recruited at those sites only; other participants were recruited through online advertisement
* Active Duty Service Members (MAMC & WPMC) and Veterans (online arm)
* Between the ages of 18-65
* English language fluency

Exclusion Criteria:

* Active psychosis or mania,
* Serious suicidal intent requiring hospitalization or immediate treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Multidimensional Assessment of Interoceptive Awareness | Within one week of completing the intervention. Also administered at one and three month follow-up.
  This 35-item scale has 8 subscales that measure the ability to recognize and accurately identify emotions and physiological sensations.

SECONDARY OUTCOMES:
Suicidal ideation | Within one week of completing the intervention. Also administered at one and three month follow-up.
  Depression Symptom Index-Suicidality Subscale; Beck Scale for Suicide Ideation

OTHER OUTCOMES:
Body Functionality | Within one week of completing the intervention. Also administered at one and three month follow-up.
  Functionality Appreciation Scale

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Wright Patterson Medical Center, Dayton, Ohio
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared with the Military Suicide Research Consortium and uploaded on a quarterly basis.

REFERENCES:
- [Background] Craig AD. How do you feel? Interoception: the sense of the physiological condition of the body. Nat Rev Neurosci. 2002 Aug;3(8):655-66. doi: 10.1038/nrn894. PMID 12154366
- [Background] Forrest LN, Smith AR, White RD, Joiner TE. (Dis)connected: An examination of interoception in individuals with suicidality. J Abnorm Psychol. 2015 Aug;124(3):754-63. doi: 10.1037/abn0000074. PMID 26147323
- [Background] Smith A, Forrest L, Velkoff E. Out of touch: Interoceptive deficits are elevated in suicide attempters with eating disorders. Eat Disord. 2018 Jan-Feb;26(1):52-65. doi: 10.1080/10640266.2018.1418243. PMID 29384458
- [Background] Guerra VS, Calhoun PS; Mid-Atlantic Mental Illness Research, Education and Clinical Center Workgroup. Examining the relation between posttraumatic stress disorder and suicidal ideation in an OEF/OIF veteran sample. J Anxiety Disord. 2011 Jan;25(1):12-8. doi: 10.1016/j.janxdis.2010.06.025. Epub 2010 Jul 7. PMID 20709493
- [Background] Nademin E, Jobes DA, Pflanz SE, Jacoby AM, Ghahramanlou-Holloway M, Campise R, Joiner T, Wagner BM, Johnson L. An investigation of interpersonal-psychological variables in air force suicides: a controlled-comparison study. Arch Suicide Res. 2008;12(4):309-26. doi: 10.1080/13811110802324847. PMID 18828034
- [Background] Shelef L, Levi-Belz Y, Fruchter E. Dissociation and acquired capability as facilitators of suicide ideation among soldiers. Crisis. 2014;35(6):388-97. doi: 10.1027/0227-5910/a000278. PMID 25231854